CLINICAL TRIAL: NCT01744535
Title: Pilot Trial of "My Meal Mate" (MMM), a Smartphone Application Designed to Facilitate Weight Loss.
Brief Title: Pilot Trial of "My Meal Mate" (MMM), a Smartphone Application for Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Michelle Carter, Research Dietitian, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G0802108
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Overweight
Keywords: smartphone; smartphone app; smartphone application; obesity; overweight; self monitoring
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Paper food diary (Active Comparator)
  Interventions: Behavioral: Paper food diary
- Online food diary (Active Comparator)
  Interventions: Behavioral: Online food diary
- "My Meal Mate" (smartphone application) (Experimental): A smartphone application called "My Meal Mate" (MMM) designed to facilitate weight loss. The app allows system users to set a goal for weight loss and self monitor diet and activity in an electronic diary. Users can select foods from the large "Weight Loss Resources" food database. Instant nutritional feedback is provided along with weekly feedback by text message.
  Interventions: Behavioral: "My Meal Mate" (smartphone application)

INTERVENTIONS:
Behavioral: "My Meal Mate" (smartphone application) — A smartphone application called "My Meal Mate" (MMM) designed to facilitate weight loss. The app allows system users to set a goal for weight loss and self monitor diet and activity in an electronic diary. Users receive instant nutritional feedback and feedback via text message.
  Arms: "My Meal Mate" (smartphone application)
Behavioral: Paper food diary — The paper food diary is provided by a commerical slimming organisation called "Weight Loss Resources". The diary allows the user to record daily food and drink consumed. It is accompanied by a book which provides a database of the nutritional content of 40,000 food and drinks. The diary also encourages participants to record their physical activity.
  Arms: Paper food diary
Behavioral: Online food diary — The online food diary is provided by a commerical slimming organisation called "Weight Loss Resources". The electronic diary allows the user to record daily food and drink consumed. System users are also encouraged to record their physical activity.
  Arms: Online food diary

SUMMARY:
The aim of this study is to implement an exploratory pilot trial of "My Meal Mate" (MMM), a smartphone application developed to facilitate weight loss, assessing its feasibility and acceptability. Overweight and obese adults will be recruited from large employers within the local area. The trial will aim to recruit a sample size of 135 which is a pragmatic decision based on randomizing 45 people to each arm. Participants will be randomized to one of three groups. The researchers have developed a smartphone application for weight loss called "My Meal Mate" (MMM) which incorporates a large branded food and drink database. MMM was developed using focus group data collected from potential system users and by benchmarking with similar commercially available diet tracking applications. One group will receive a smartphone with the MMM app downloaded on it, one group will receive access to an online food diary and one group will be given a paper food diary. Participants will be asked to set a goal for weight loss and self-monitor their food intake and activity using their allocated study equipment. Participants will be weighed at the beginning of the trial, at 6 weeks and at 6 months. Feasibility and acceptability outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* BMI equal to or greater than 27 kg/m2
* Willing to commit the necessary time and effort to the study,
* Employed by a large employer in Leeds (and expects to continue to be employed there for the next 12 months),
* Able to read and write in English,
* Able to access the internet,
* Willing to be randomised to one of three groups.

Exclusion Criteria:

* Pregnant, planning a pregnancy within next 12 months, lactating
* Has had surgery for weight loss
* Taking the medication sertraline (due to associations with weight gain)
* Taking anti-obesity medications or medications for diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Adherence to the trial | 6 months
  The number of completers in each group is a feasibility outcome.
Adherence to the intervention arms | 6 months
  The number of days with a plausible record of diet (>500-5000 kcal recorded) in each arm is a feasibility outcome.

SECONDARY OUTCOMES:
Weight change (kg) | 6 months
  Weight (kg) has been objectively measured at baseline and 6 months.
BMI change | 6 months
  BMI(kg/m2) has been objectively measured at baseline and 6 months.
change in body fat percentage | 6 months
  Body fat (%) has been objectively measured at baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Cade, Professor, Principal Investigator — University of Leeds
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Background] Carter MC, Burley VJ, Nykjaer C, Cade JE. 'My Meal Mate' (MMM): validation of the diet measures captured on a smartphone application to facilitate weight loss. Br J Nutr. 2013 Feb 14;109(3):539-46. doi: 10.1017/S0007114512001353. Epub 2012 May 3. PMID 22717334
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Carter MC, Burley VJ, Cade JE. Weight Loss Associated With Different Patterns of Self-Monitoring Using the Mobile Phone App My Meal Mate. JMIR Mhealth Uhealth. 2017 Feb 2;5(2):e8. doi: 10.2196/mhealth.4520. PMID 28153814
- [Derived] Carter MC, Burley VJ, Nykjaer C, Cade JE. Adherence to a smartphone application for weight loss compared to website and paper diary: pilot randomized controlled trial. J Med Internet Res. 2013 Apr 15;15(4):e32. doi: 10.2196/jmir.2283. PMID 23587561